CLINICAL TRIAL: NCT03776604
Title: Multi-center, Open, One-arm Clinical Study Evaluating the Efficacy and Safety of Jinyouli (PEGylated Recombinant Human Granulocyte Stimulating Factor, PEG-rhG-CSF) in Preventing Neutropenia After Chemotherapy in Elderly Patients With Small Cell Lung Cancer
Brief Title: PEG-rhG-CSF in Elderly Patients With Small Cell Lung Cancer Receiving Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-JYL-SCLC-01
Record Dates: First submitted 2018-12-10; First posted 2018-12-17 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Small Cell Lung Cancer; PEG-rhG-CSF
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Intervention Model Description: Subjects with newly diagnosed small cell lung cancer who met the inclusion/exclusion criteria were prophylactically administered the test drug PEG-rhG-CSF 48 h after chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEG-rhG-CSF (Experimental): Jin Youli(PEG-rhG-CSF): The dose is determined according to the patient's weight. Those who weighed more than ≥45kg were given 6mg/time, and those who were <45kg or less were given 3mg/time. Administration method: Subcutaneous injection, the lower edge of the deltoid muscle of both arms is preferentially selected, and each injection is injected once every chemotherapy cycle.
  Dosing time: 48 h after chemotherapy.
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — Subjects with newly diagnosed small cell lung cancer who met the inclusion/exclusion criteria were prophylactically administered the test drug PEG-rhG-CSF 48 h after chemotherapy.
  Jin Youli（PEG-rhG-CSF）: The dose is determined according to the patient's weight. Those who weighed more than ≥45kg were given 6mg/time, and those who were <45kg or less were given 3mg/time. Administration method: Subcutaneous injection, the lower edge of the deltoid muscle of both arms is preferentially selected, and each injection is injected once every chemotherapy cycle.
  Dosing time: 48 h after chemotherapy.

SUMMARY:
Evaluation of the efficacy and safety of Jinyouli in preventing neutropenia in multiple chemotherapy cycles in elderly patients with small cell lung cancer through a multicenter, open, one-arm study Subjects with newly diagnosed small cell lung cancer who met the inclusion/exclusion criteria, chemotherapy regimen: etoposide: 100 mg/m2, d1-3, carboplatin: AUC=5, d1, q21d, prophylactic use test 48 h after chemotherapy Drug PEG-rhG-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years old, gender is not limited;
* Small cell lung cancer patients diagnosed by histopathology or cytology;
* ECOG = 0-1;
* The estimated survival period is more than 3 months;
* No obvious signs of hematological disease, defined as Hb≥90g/dL, WBC≥4.0×10^9/L, ANC≥2×10^9/L, PLT≥100×10^9/L before enrollment. And no bleeding tendency;
* No obvious abnormalities were observed in the electrocardiogram examination;
* Liver function tests ALT, AST, TBIL indicators are within 2.5 times the upper limit of normal values. If due to liver metastasis, the above indicators should be within 5 times of the upper limit of normal. If LDH is elevated due to non-tumor causes, LDH should be ≤ 2.5 times the upper limit of normal; if LDH is elevated due to tumor, it can be enrolled;
* Renal function test BUN, UA within 1.5 times the upper limit of normal value, creatinine clearance rate> 60ml / min;
* Subjects (or their legal representatives/guardians) must sign an informed consent form indicating that they understand the purpose of the study, understand the necessary procedures for the study, and are willing to participate in the study.

Exclusion Criteria:

* There are currently uncontrollable infections, body temperature ≥ 38.0 ° C;
* Patients with previous malignant tumors that have not been cured or have bone marrow metastasis;
* Patients with prophylactic antibiotics;
* Accepting other test drugs at the same time or participating in other clinical trials;
* Those who are allergic to this product or other genetically engineered E. coli-derived biological products;
* The patient has any myelodysplastic and other blood system diseases;
* Patients who have received hematopoietic stem cell transplantation or organ transplantation;
* The patient has a severe mental or neurological condition that affects informed consent and/or adverse reaction presentation or observation.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade III/IV neutropenia in the first cycle of PEG-rhG-CSF. | through first cycle of PEG-rhG-CSF,an average of 1 month
  The incidence of grade III/IV neutropenia in the first cycle of PEG-rhG-CSF.
The incidence of grade III/IV neutropenia in the second cycle of PEG-rhG-CSF. | through second cycle of PEG-rhG-CSF,an average of 1 month
  The incidence of grade III/IV neutropenia in the second cycle of PEG-rhG-CSF.

SECONDARY OUTCOMES:
The incidence of febrile neutropenia in cycles 1 and 2 | through 1-2 cycles of PEG-rhG-CSF,an average of 2 month
  Febrile neutropenia (FN) is defined as oral temperature >38.3 ° C (underarm temperature >38.1 ° C) or continuous measurement of oral temperature >38 ° C (underarm temperature >37.8 ° C) in 2 h, and ANC <0.5×10^9/L, or expected to be <0.5×10^9/L
The ANC recovery time in cycles 1 and 2 | through 1-2 cycles of PEG-rhG-CSF,an average of 2 month
  Defined as the patients who appear ANC<2.0×10^9/L，from the first day of chemotherapy, to the time of ANC≥ 2.0×10^9/L, take the median.
The incidence of infection | up to 30 days after the patient study completion
The incidence of antibiotic use | up to 30 days after the patient study completion
Incidence of chemotherapy dose adjustment due to neutropenia | through the study completion,an average of 3 months
Chemotherapy delay time | through the study completion,an average of 3 months
Incidence of chemotherapy delay caused by neutropenia | through the study completion,an average of 3 months
The duration of febrile neutropenia in cycles 1 and 2 | through 1-2 cycles of PEG-rhG-CSF,an average of 2 month

OTHER OUTCOMES:
Incidence and severity of adverse events | through the study completion,an average of 3 months
  All adverse events will be recorded from the time of signing the informed consent form to 30 days after the last dose. Adverse events 30 days after the last dose, only those adverse events associated with the study drug were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Bejing Cancer Hospital, Beijing, Beijing Municipality, China